CLINICAL TRIAL: NCT05758675
Title: Study on the Antibody Level Against SARS-CoV-2 in Dazhu County in 2023
Brief Title: Study on the Antibody Level Against SARS-CoV-2 （COVID-19）in Dazhu County in 2023
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCT-Dazhu-Screening-1
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ≥ 60 years old population: around 2000 subjects will be screened.
- 18~59 years old population: around 3000 subjects will be screened.
- < 18 years old: around 15000 subjects will be screened.

SUMMARY:
About 15,000 to 25,000 subjects will be screened. Their information will be collected, venous blood will be sampled, their serum antibody levels will be detected, and the incidence of COVID-19 wil be followed up.

DETAILED DESCRIPTION:
Data of the following will be collected:

1. Demographic data,including Name, Gender, Ethnic groups, ID Card number (age automatically calculated), Height/weight (automatic BMI calculation);
2. Previous disease/surgical history; 3. Previous COVID-19 infections; 4. COVID-19 vaccination history; 5. Infection after this screening; 6. Screening information for COVID-19 antibodies.

Atibody level against SARS-CoV-2 will be test.

ELIGIBILITY:
Inclusion Criteria:

* The age when signing ICF should be ≥3 year, male or female.
* The Subject and/or guardian or client of both parties are able to sign a written ICF and voluntarily participate in the trial, fully understand the trial procedure, the risks of participating in the study.
* Healthy subjects or subjects with stable underlying diseases. Stable underlying diseases were defined as those who were in stable condition at least 3 months before inclusion in the study, had no significant change in treatment regimen and had not been admitted to hospital due to disease progression.

Exclusion Criteria:

* a history of contraindications for venous blood collection such as thrombocytopenia or other clotting disorders.
* Current severe or uncontrollable cardiovascular disease, endocrine disease, blood and lymphatic system disease, liver and kidney disease, respiratory system disease, metabolic and skeletal system disease, or malignancy.
* If it is not in line with the benefit maximization of the subjects, the investigator determines that it is not suitable to participate in clinical research.

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Screening by sampling from natural communities.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of antibody against SARS-CoV-2 | From Day 0 to Day 180
  Concentration of antibody against SARS-CoV-2 in different age groups

SECONDARY OUTCOMES:
Relation between collected information and antibody concentration | From Day 0 to Day 180
  Analysis of the correlation between the antibody level and the collected information.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhou, M.D., Principal Investigator — Dazhu County Center for Disease Control and Prevention
Locations (1):
- Dazhu County Center for Disease Control and Prevention, Dazhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Distribution analysis and correlation analysis of antibody will be done and published in academic journals.